CLINICAL TRIAL: NCT01140633
Title: Novel Measures and Theory of Pediatric Antiretroviral Therapy Adherence in Uganda
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Jessica Haberer, MD, Assistant in Medicine, Massachusetts General Hospital
Other Study IDs: 2009-P-001062; K23MH087228 (NIH)
Record Dates: First submitted 2010-06-07; First posted 2010-06-09 (Estimated); Last update posted 2013-09-02 (Estimated); Status verified 2013-08

CONDITIONS: HIV-infection/Aids
Keywords: HIV/AIDS; pediatric; wireless adherence monitoring; HIV Infections
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples with HIV viral DNA.
Oversight: Data Monitoring Committee: No

SUMMARY:
Current measures of adherence detect problems weeks to months after they occur. Because the HIV virus rapidly begins replicating and mutating in the absence of effective antiretroviral therapy, treatment failure may develop before an intervention can be deployed. Real-time objective adherence monitoring could redirect efforts from a reactive response to the proactive prevention of treatment failure. Because adherence is so closely associated with viral suppression, accurate adherence monitoring could also strategically limit viral monitoring only to those patients at a defined risk for viral rebound.

This observational study is assessing a wireless adherence monitoring device and mobile phone-based adherence data collection among caregivers of children under the age of ten years in Mbarara, Uganda. It involves both quantitative and qualitative measures of the feasibility and acceptability of these measures, as well as circumstances of adherence lapses and other individual and cultural factors affecting adherence. The qualitative data will be used to explore models of adherence behavior, which will likely include the child-caregiver dynamic, the child's mental and physical health, and social support mechanism.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

* age 1 to 10 years
* HIV-infected, meeting Ugandan criteria for antiretroviral therapy
* living within 30 km of Mbarara, Uganda

Exclusion Criteria:

* lack of mobile-phone reception

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: young children receiving HIV antiretroviral therapy in a rural African setting
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-04; Primary Completion 2011-01 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Distribution of adherence | Monthly adherence levels will be determined over the six-month study period.
  Distribution of adherence based on wireless adherence monitoring devices and interactive voice response (IVR) or short message service (SMS) self report by caregivers of HIV-infected children under ten years old in Mbarara, Uganda.

SECONDARY OUTCOMES:
Feasibility and acceptability of wireless adherence measures | Assessments will be made a the one-month time point.
  Quantitive rating and qualitative description of the feasibility and acceptability of wireless adherence measures
Model of adherence behavior | Data collected at baseline and during adherence interruptions will be analyzed at the end of the six-month study period.
  Qualitative data will be used to explore a theoretical model of adherence behavior among young children in a rural African setting

CONTACTS AND LOCATIONS:
Overall Officials: Jessica E Haberer, MD, MS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mbarara University Teaching Hospital, Mbarara, Uganda